CLINICAL TRIAL: NCT05237830
Title: Effectiveness of Intraoperative Cell Salvage in Aseptic Revision Total Hip Arthroplasty: a Single-center Retrospective Study
Brief Title: Effectiveness of Intraoperative Cell Salvage in Aseptic Revision Total Hip Arthroplasty.
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Michele Carella, Principal Investigator, University of Liege
Other Study IDs: Cell-salvage
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Revision of Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Use: Patients in whom the cell saver was effectively used
  Interventions: Procedure: Use of Cell Salvage in revision of total hip arthroplasty
- Not Use: Patients in whom the cell saver wasn't effectively used
  Interventions: Procedure: Use of Cell Salvage in revision of total hip arthroplasty

INTERVENTIONS:
Procedure: Use of Cell Salvage in revision of total hip arthroplasty — The effective use of the cell saver was defined as the ability to re-transfuse at least 125 mL of re-suspended red blood cells with a hematocrit of 60 %.

SUMMARY:
Intraoperative cell salvage is an important measure of patient blood management but its effectiveness in patients undergoing revision total hip arthroplasty remains unclear. Over the last decade, we have used intraoperative cell salvage systematically in this group of patients. However, since the use of cell salvage has a cost and requires additional resources, we decided to retrospectively investigate its usefulness in this particular indication.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were adults undergoing elective aseptic revision of hip arthroplasty at the department of orthopedic surgery of the University Hospital of Liege between 01 January 2011 and 31 December 2020.

Exclusion Criteria:

* Patients undergoing revision for infection or with local malignancies were excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Revision of arthroplasty was defined as the exchange of any component of the hip prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Cell savage use | during the surgical procedure
  The primary outcome was the proportion of patients in whom the cell saver was effectively used (%)

SECONDARY OUTCOMES:
Re-infused | during the surgical procedure
  Total volume of re-suspended blood re-infused (mL)
Hemoglobin | during the surgical procedure
  Post-operative hemoglobin level (g/dL)
Allogenic Transfusion | 7 days
  The need for allogenic blood transfusion (unit)
Aspirated blood | during the surgical procedure
  The total volume of blood aspirated into the reservoir (mL)
Fluid | during the surgical procedure
  The total amount of fluid infused (mL)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenky M, Shaner J, Rasouli MR, Han SB, Parvizi J, Hozack WJ. Intraoperative blood salvage in revision total hip arthroplasty: who benefits most? J Arthroplasty. 2014 Jun;29(6):1298-300. doi: 10.1016/j.arth.2013.12.009. Epub 2013 Dec 14. PMID 24412146
- [Background] Palmer AJR, Lloyd TD, Gibbs VN, Shah A, Dhiman P, Booth R, Murphy MF, Taylor AH, Kendrick BJL; collaborators. The role of intra-operative cell salvage in patient blood management for revision hip arthroplasty: a prospective cohort study. Anaesthesia. 2020 Apr;75(4):479-486. doi: 10.1111/anae.14989. Epub 2020 Feb 9. PMID 32037522
- [Background] Rigal JC, Riche VP, Tching-Sin M, Fronteau C, Huon JF, Cadiet J, Boukhari R, Vourc'h M, Rozec B. Cost of red blood cell transfusion; evaluation in a French academic hospital. Transfus Clin Biol. 2020 Nov;27(4):222-228. doi: 10.1016/j.tracli.2020.08.002. Epub 2020 Aug 15. PMID 32810606
- [Background] Goel R, Patel EU, Cushing MM, Frank SM, Ness PM, Takemoto CM, Vasovic LV, Sheth S, Nellis ME, Shaz B, Tobian AAR. Association of Perioperative Red Blood Cell Transfusions With Venous Thromboembolism in a North American Registry. JAMA Surg. 2018 Sep 1;153(9):826-833. doi: 10.1001/jamasurg.2018.1565. PMID 29898202
- [Background] Walsh TS, Palmer J, Watson D, Biggin K, Seretny M, Davidson H, Harkness M, Hay A. Multicentre cohort study of red blood cell use for revision hip arthroplasty and factors associated with greater risk of allogeneic blood transfusion. Br J Anaesth. 2012 Jan;108(1):63-71. doi: 10.1093/bja/aer326. Epub 2011 Oct 27. PMID 22037224